CLINICAL TRIAL: NCT05446324
Title: SENtinel Lymph Node Mapping With GAllium-68-tilmanocept PET/CT in High/High-intermediate Risk Endometrial Cancer: a Pilot Study
Brief Title: Feasibility of Gallium-68-tilmanocept PET/CT for Sentinel Lymph Node Detection in Endometrial Cancer
Acronym: SENGA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Ronald Zweemer, Prof. dr. Ronald P. Zweemer, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL81058.041.22
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Sentinel lymph node mapping; Image guided surgery
MeSH Terms: conditions — Endometrial Neoplasms | interventions — gallium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-tilmanocept PET/CT (Experimental): All participants receive 68Ga-tilmanocept PET/CT imaging in adjunct to standard-of-care (SLN mapping with intraoperative ICG).
  Interventions: Drug: Gallium-68-tilmanocept

INTERVENTIONS:
Drug: Gallium-68-tilmanocept — All participants receive a cervical injection with 10 MBq 68Ga-tilmanocept in an outpatient setting (at least one week) before surgery. Within 30-90 minutes post-injection a PET with contrast enhanced CT is performed (PET/CT). Data (i.e. detection rate) from the imaging modalities are collected.
  Other Names: 68Ga-tilmanocept

SUMMARY:
This pilot study evaluates the feasibility of 68Ga-tilmanocept PET/CT for SLN mapping in patients with endometrial cancer.

DETAILED DESCRIPTION:
Rationale: Currently, the use of indocyanine green (ICG) is the most widely accepted sentinel lymph node (SLN) mapping technique in endometrial cancer but the acquired SLN detection rates greatly vary. We propose that adding preoperative imaging with the radiotracer Gallium-68-tilmanocept (68Ga-tilmanocept) PET/CT can further improve SLN mapping in patients with endometrial cancer and reliably guide the surgeon towards the true SLN intraoperatively.

Objective: To evaluate the feasibility of sentinel lymph node imaging with 68Ga-tilmanocept PET/CT.

Study design: Non-randomised, single-centre, single-arm pilot study in the UMC Utrecht.

Study population: Patients with clinically stage I-II high/high-intermediate risk endometrial cancer scheduled for robot-assisted pelvic and para-aortic lymphatic staging (including SLN procedure). A total of 10 patients will be included.

Intervention (if applicable): Preoperative cervical injection of 68Ga-tilmanocept followed by preoperative PET/CT imaging (in adjunct to the standard-of-care: intraoperative injection with indocyanine green (ICG) with real-time near-infrared (NIR) fluorescence imaging). Injection of 68Ga-tilmanocept is performed by the gynaecologist in an outpatient setting. The PET/CT (PET + contrast enhanced CT abdomen) will be performed 30-90 minutes after tracer injection.

Main study parameters/endpoints: Feasibility of 68Ga-tilmanocept PET/CT for SLN mapping, which is evaluated by its SLN detection rate.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Extra burden for subjects concerns an additional site visit for cervical injection followed by PET/CT imaging with a total duration of two hours (including waiting time of ~60 minutes). The preoperative injection with 68Ga-tilmanocept while patient is awake adds minimal discomfort to the patient. The extra administration of 10 MBq 68Ga-tilmanocept followed by PET/CT, resulting in a radiation of 6.3 mSv, is considered an acceptable radiation burden to the subjects. Adverse reactions after injection of radiolabelled tilmanocept rarely occur. No additional blood samples, follow-up visits or physical examinations are needed during this study. The additional site visit does not delay the scheduled standard care.

Subjects may benefit from this study since the SLN detection rate could be increased and/or faster by adding 68Ga-tilmanocept PET/CT to the diagnostic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical FIGO 2012 stage I-II high/high-intermediate risk endometrial cancer;
* Scheduled for robot-assisted full pelvic and para-aortic staging;
* Age ≥18 years and able to provide informed consent.

Exclusion Criteria:

* Pregnancy or current breastfeeding;
* Prior severe allergic reaction to iodine;
* Severe renal insufficiency (stage 3 or 4);
* Clinical or radiological evidence of metastatic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of 68Ga-tilmanocept PET/CT for SLN mapping | One week post-PET/CT
  Assessed by the SLN detection rate with 68Ga-tilmanocept PET/CT. Overall SLN detection rate is defined as the proportion of patients in which at least one SLN is detected. Bilateral SLN detection rate is defined as the proportion of patients with at least one SLN detected in each hemipelvis or para-aortic side.

SECONDARY OUTCOMES:
Correlation between SLN detection rate and anatomical location with preoperative 68Ga-tilmanocept PET/CT versus intraoperative ICG with near-infrared fluorescence. | Intraoperative
  Preoperative and intraoperative localisation of the detected SLNs will be reported according to a fixed format.
Pathological status of SLNs | One week post-surgery
  Assessed as: tumour negative, macrometastasis (diameter >2.0 mm), micrometastasis (diameter between 0.2 and 2.0 mm) or isolated tumour cells (diameter <0.2 mm or individual tumour cells).
Adverse events related to SLN mapping with 68Ga-tilmanocept PET/CT | Up to one hour post-PET/CT
  Graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis G Gerestein, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Cornelis G Gerestein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No